CLINICAL TRIAL: NCT01744379
Title: A Phase 1, Randomized, Double-Blind, Placebo-Controlled Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Pharmacodynamics of Single and Multiple Doses of Lesinurad in Healthy Male Japanese Subjects
Brief Title: Single and Multiple Dose Study in Japanese
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: Ardea Biosciences, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: RDEA594-125
Record Dates: First submitted 2012-11-29; First posted 2012-12-06 (Estimated); Last update posted 2013-06-19 (Estimated); Status verified 2013-06

CONDITIONS: Gout
MeSH Terms: conditions — Gout | interventions — lesinurad

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (5):
- 200 mg lesinurad (Experimental): 200 mg lesinurad or placebo fasted and fed
  Interventions: Drug: Lesinurad; Drug: Placebo
- 400 mg lesinurad (Experimental): 400 mg lesinurad or placebo fasted and fed
  Interventions: Drug: Lesinurad; Drug: Placebo
- 100 mg lesinurad (Experimental): 100 mg lesinurad or placebo fasted and fed
  Interventions: Drug: Lesinurad; Drug: Placebo
- 50 mg lesinurad (Experimental): 50 mg lesinurad or placebo fasted and fed
  Interventions: Drug: Lesinurad; Drug: Placebo
- 600 mg lesinurad (Experimental): 600 mg lesinurad or placebo fasted and fed
  Interventions: Drug: Lesinurad; Drug: Placebo

INTERVENTIONS:
Drug: Lesinurad
Drug: Placebo

SUMMARY:
This study will explore the safety, tolerability, and serum uric acid lowering effect of lesinurad in healthy Japanese males to allow comparison with the Western population.

DETAILED DESCRIPTION:
While there is extensive clinical experience with lesinurad in the Western population, it is recognized that both intrinsic and extrinsic factors may impact the PK, PD, safety, and dose response in different ethnic populations. The purpose of this study is to explore the safety, tolerability, pharmacokinetic (PK), and pharmacodynamic (PD) of single and multiple doses of lesinurad in healthy Japanese males, and to allow comparison of these parameters with the Western population.

ELIGIBILITY:
Inclusion Criteria:

* Able to understand the study procedures, the risks involved and willing to provide written Informed Consent before the first study related activity.
* Healthy adult subjects born in Japan
* All laboratory parameters should be within normal limits or considered not clinically significant by the investigator.
* Screening serum uric acid level >= 4.5 mg/dL.
* Subjects must be free of any clinically significant disease that requires a physician's care and/or would interfere with study evaluations or procedures.
* Subject does not have clinically relevant abnormalities in blood pressure, heart rate, body temperature, and respiratory rate, as per the Investigator's judgment.

Exclusion Criteria:

* Positive serology to Human Immunodeficiency Virus (HIV-1 and HIV-2).
* Positive test for active Hepatitis B or Hepatitis C infection.
* History of kidney stones.
* Undergone major surgery within 3 months of Day 1.
* Subject has received the last dose of an investigational drug (or treatment with a medical device) within 30 days or 5 half-lives (whichever is longer) of the investigational drug prior to Day 1 or are currently participating in another study of an investigational drug (or medical device).
* Prior exposure to lesinurad (RDEA594) or RDEA806.

Ages: 20 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-12; Primary Completion 2013-03 (Actual); Study Completion 2013-05 (Actual)

PRIMARY OUTCOMES:
Incidence of Adverse Events and Changes in Laboratory Parameters | 5 to 6 weeks
Pharmacokinetic (PK) profile of lesinurad from plasma and urine in terms of AUC, tmax, cmax and t1/2. | Day -1 through 12
  AUC: area under the plasma concentration time curve from zero to 24 hours post dose and from zero to infinity; tmax: time to maximum plasma concentration; cmax: maximum observed plasma concentration t1/2: terminal elimination half life
Pharmacodynamic (PD) profile of lesinurad from serum and urine in terms of sUA concentration, renal clearance, urine uric acid excretion, and fractional excretion. | Day 1 through 12

CONTACTS AND LOCATIONS:
Overall Officials: S Bradley, MD, Study Director — Ardea Biosciences, Inc.
Locations (1):
- Glendale, California, United States